CLINICAL TRIAL: NCT06693726
Title: ANGIOtensin II for Septic Shock in the Emergency Department: ANGIO-ED Study
Brief Title: Early Angiotensin II in the Emergency Department
Acronym: ANGIO-ED
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Brett A Faine (Other)
Responsible Party: Sponsor-Investigator, Brett A Faine, Clinical Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202406277
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Septic Shock
Keywords: Angiotensin II
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Angiotensin II Infusion (Experimental)
  Interventions: Drug: Angiotensin II Infusion

INTERVENTIONS:
Drug: Angiotensin II Infusion — Angiotensin II continuous infusion

SUMMARY:
This pilot study will enroll 20 patients with septic shock and require emergent vasopressor support in the emergency department (ED). The primary objective of the study is to determine the feasibility of early peripheral administration of angiotensin II for treatment of septic shock in the ED

DETAILED DESCRIPTION:
Following informed consent, patients will receive intravenous angiotensin II (AT-II) infusion for blood pressure support. The patient will remain on the AT-II infusion for 60 minutes prior to determining patient response which will be determined by recording the concurrent dose of norepinephrine and MAP every 10 minutes from initiation. If a positive response (e.g., norepinephrine dose reduction) is witnessed, the AT-II infusion will be titrated off after a maximum of 6 hours or when infusion is completed, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥18; and
2. Requiring norepinephrine at a dose of 0.05-0.25 mcg/kg/min mcg/kg/minute despite adequate fluid resuscitation; and
3. Receiving intravenous antibiotics or clinician's intention to administer antibiotics at the time of enrollment; and
4. Can provide written informed consent (or legally authorized representative).

Exclusion Criteria

1. Acute coronary syndrome;
2. Cardiogenic shock;
3. Patients with a history of mesenteric ischemia;
4. Patients with a history of having an aortic dissection or abdominal aortic aneurysm;
5. Patients with an expected lifespan of <12 hours;
6. Patients with hemorrhagic shock (e.g., actively receiving transfusion of packed red blood cells);
7. Active administration of two vasoactive agents before enrollment; and
8. Pre-existing thromboembolic disease or inability to tolerate pharmacologic VTE prophylaxis.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of completing all clinical trial activities | From enrollment to the end of treatment up to 6 hours after the angiotensin II infusion is initiated
  Percentage of patients who provide informed consent and receive angiotensin II infusion in the emergency department

SECONDARY OUTCOMES:
Mean arterial pressure response | 60 minutes after the intiation of angiotensin II infusion
  Change in mean arterial pressure
Mean norepinephrine dose (during angiotensin II infusion) | 60 minutes after the intiation of angiotensin II infusion
  Change in norepinephrine dose (mcg/kg/minute) after the initiation of angiotensin II infusion
Mean norepinephrine dose (post angiotensin II infusion) | 60 minutes after the completion of the angiotensin II infusion
  Mean norepinephrine dose (mcg/kg/minute) after the completion of the angiotensin II infusion

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the manuscript, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, CSR
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] Khanna A, English SW, Wang XS, Ham K, Tumlin J, Szerlip H, Busse LW, Altaweel L, Albertson TE, Mackey C, McCurdy MT, Boldt DW, Chock S, Young PJ, Krell K, Wunderink RG, Ostermann M, Murugan R, Gong MN, Panwar R, Hastbacka J, Favory R, Venkatesh B, Thompson BT, Bellomo R, Jensen J, Kroll S, Chawla LS, Tidmarsh GF, Deane AM; ATHOS-3 Investigators. Angiotensin II for the Treatment of Vasodilatory Shock. N Engl J Med. 2017 Aug 3;377(5):419-430. doi: 10.1056/NEJMoa1704154. Epub 2017 May 21. PMID 28528561
- [Background] Chawla LS, Busse L, Brasha-Mitchell E, Davison D, Honiq J, Alotaibi Z, Seneff MG. Intravenous angiotensin II for the treatment of high-output shock (ATHOS trial): a pilot study. Crit Care. 2014 Oct 6;18(5):534. doi: 10.1186/s13054-014-0534-9. PMID 25286986
- [Background] Wieruszewski PM, Bellomo R, Busse LW, Ham KR, Zarbock A, Khanna AK, Deane AM, Ostermann M, Wunderink RG, Boldt DW, Kroll S, Greenfeld CR, Hodges T, Chow JH; Angiotensin II for the Treatment of High-Output Shock 3 (ATHOS-3) Investigators. Initiating angiotensin II at lower vasopressor doses in vasodilatory shock: an exploratory post-hoc analysis of the ATHOS-3 clinical trial. Crit Care. 2023 May 5;27(1):175. doi: 10.1186/s13054-023-04446-1. PMID 37147690
- [Background] Avni T, Lador A, Lev S, Leibovici L, Paul M, Grossman A. Vasopressors for the Treatment of Septic Shock: Systematic Review and Meta-Analysis. PLoS One. 2015 Aug 3;10(8):e0129305. doi: 10.1371/journal.pone.0129305. eCollection 2015. PMID 26237037